CLINICAL TRIAL: NCT05515471
Title: A Phase 3, Multi-Center, Randomized, Double-Masked, Saline-Controlled Trial to Evaluate the Effect of SHR8058 on Signs and Symptoms of Dry Eye Disease Associated With Meibomian Gland Dysfunction
Brief Title: Effect of SHR8058 on Signs and Symptoms of Dry Eye Disease Associated With Meibomian Gland Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHR8058-301
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Treatment of Dry Eye Disease With Meibomian Gland Dysfunction

STUDY DESIGN:
Intervention Model Description: SHR8058 eye drops compared with placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A: SHR8058 eye drops (Experimental)
  Interventions: Drug: SHR8058 eye drops
- Treatment group B: saline eye drops (Placebo Comparator)
  Interventions: Drug: saline eye drops.

INTERVENTIONS:
Drug: SHR8058 eye drops — SHR8058 eye drops
  Arms: Treatment group A: SHR8058 eye drops
Drug: saline eye drops. — saline eye drops.
  Arms: Treatment group B: saline eye drops

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of SHR8058 eye drops for patients with dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

1. Signed ICF (Informed Consent Form)
2. Subject-reported history of Drye Eye Disease (DED) in both eyes
3. Ability and willingness to follow instructions, including participation in all study assessments and visits

Exclusion Criteria:

1. clinically significant slit lamp findings or abnormal lid anatomy at screening, including eye trauma, pterygium, active blepharitis, and active lid margin inflammation;
2. Stevens-Johnson syndrome or other severe systemic autoimmune diseases;
3. underwent LipiFlow procedure or intention pulsed light therapy within 6 months before baseline, or received Meibomian gland massage treatment within 2 weeks before baseline;
4. received or removed permanent lacrimal plug within 3 months before baseline;
5. DED secondary to scarring, radiation, alkali burns, cicatricial pemphigoid, or destruction of conjunctival goblet cells;
6. ocular or periocular malignancy;
7. active ocular allergies, or allergy to the study drug or its components;
8. ongoing ocular or systemic infection;
9. use of contact lenses within 1 month before screening;
10. intraocular surgery or ocular laser surgery within 6 months before enrollment;
11. uncontrolled systemic disease or history of herpetic keratitis;
12. use of topical steroids, topical cyclosporine, lifitegrast, serum tears, or topical anti-glaucoma medication within 60 days before screening;
13. used any known oral drugs that could have caused eye dryness within 1 month before screening;
14. participated in or were participating in other clinical trials drugs or device within 60 days before baseline;
15. inappropriate to participate for other reasons judged by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total Corneal Fluorescein Staining (NEI scale) at Day 57 | Baseline, Day 57
  The National Eye Institute (NEI) scale relies on a chart that divides the cornea into five sections (central, superior, temporal, nasal, and inferior) and assigns a value from 0 (absent) to 3 (severe) to each section, based on the amount, size, and confluence of the punctate keratitis, for a maximum total score of 15 points (sum of scores for each section).
Change from baseline in Dryness Score (visual analogue scale [VAS] Severity of Dryness) at Day 57 | Baseline, Day 57
  Study staff will ask participants to rate their severity of ocular dryness (both eyes simultaneously) by placing a vertical mark on a horizontal line to indicate the level of discomfort (0 corresponds to "no dryness" and 100% corresponds to "maximal dryness").

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhu Y, Xie J, Shi X, Sun Y. Perfluorohexyloctane Eye Drops in Premenopausal and Postmenopausal Women with Dry Eye Disease Associated with Meibomian Gland Dysfunction: A Post Hoc Analysis of a Phase 3 Trial. Curr Eye Res. 2025 Sep 2:1-7. doi: 10.1080/02713683.2025.2549289. Online ahead of print. PMID 40898391
- [Derived] Tian L, Gao Z, Zhu L, Shi X, Zhao S, Gu H, Xu G, Wang L, Dai H, Zhang H, Jin X, Ma K, Xu Y, Ma L, Pei C, Ke B, Krosser S, Zhang Y, Jie Y. Perfluorohexyloctane Eye Drops for Dry Eye Disease Associated With Meibomian Gland Dysfunction in Chinese Patients: A Randomized Clinical Trial. JAMA Ophthalmol. 2023 Apr 1;141(4):385-392. doi: 10.1001/jamaophthalmol.2023.0270. PMID 36929413